CLINICAL TRIAL: NCT02778659
Title: The Effect of Acute Hypnotic Intake Before a Night at High Altitude on Cognitive and Motor Performances
Brief Title: Hypnotic Intake and Motor and Cognitive Performances at High Altitude
Acronym: CHAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Expertise sur l'Altitude EXALT (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: CHAM
Record Dates: First submitted 2016-05-18; First posted 2016-05-20 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Physiology
MeSH Terms: interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Zolpidem Normoxia (Experimental): Acute zolpidem intake at sea level
  Interventions: Drug: Zolpidem
- Placebo Normoxia (Sham Comparator): Acute placebo intake at sea level
  Interventions: Drug: Placebo
- Zolpidem Hypoxia (Experimental): Acute zolpidem intake at high altitude
  Interventions: Drug: Zolpidem
- Placebo Hypoxia (Sham Comparator): Acute placebo intake at high altitude
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zolpidem — The hypnotic will be administrated orally at 22:00 in the evening before a sleep recording and an early wake-up at 01:00 for cognitive and motor assessment.
  Arms: Zolpidem Hypoxia; Zolpidem Normoxia
Drug: Placebo — The placebo will be administrated orally at 22:00 in the evening before a sleep recording and an early wake-up at 01:00 for cognitive and motor assessment.
  Arms: Placebo Hypoxia; Placebo Normoxia

SUMMARY:
This study aims to determine the effect of acute hypnotic intake (Zolpidem) on sleep, cognitive and motor performances and on acute mountain sickness symptoms at high altitude. Healthy subjects will be evaluated on 4 occasions (twice at sea level and twice at high altitude), after hypnotic or placebo intake. Following an early wake-up (01:00), symptoms, cognitive and motor performances will be assessed to determine potential residual effects of Zolpidem within such conditions.

ELIGIBILITY:
Inclusion Criteria:

* No sojourn above 2500 m during the past 2 months
* Coffee intake < 3 cups per day
* Non-smoker

Exclusion Criteria:

* Respiratory, cardiovascular, metabolic or neuromuscular diseases
* Psychiatric disorders
* Use of hypnotics within the past year
* Dependence syndrome (alcool, drugs, etc)
* Severe insomnia or somnolence

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2016-05; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Cognitive performance assessed using Simon cognitive test | 4 hours after drug/placebo intake
  Simon cognitive test

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Bouzat, MD PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Grenoble University Hospital, Grenoble, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No